CLINICAL TRIAL: NCT00867776
Title: Creating African-American Wellness Through Exercise: Community Driven Strategies to Improve Health
Brief Title: Creating African-American Wellness Through Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We decided to alter the intervention.
Sponsor: Oregon Health and Science University (Other)
Collaborators: African American Health Coalition (Industry)
Responsible Party: Principal Investigator, Christina M. Nicolaidis, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00005105
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Depression
Keywords: Depression; African Americans; Exercise; Culturally tailored intervention; Health disparities
MeSH Terms: conditions — Depression; Motor Activity | interventions — Self-Help Groups; Self Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AAHC Excercise Program Support Group (Experimental): Participants taking part in the AAHC Exercise Program Support Group (the intervention).
  Interventions: Behavioral: AAHC Exercise Program Support Group

INTERVENTIONS:
Behavioral: AAHC Exercise Program Support Group — 6-week community-based, culturally tailored support group program, focusing on exercise and healthy lifestyle habits. Groups will also include basic psychoeducation about depression and depression care. Groups will have up to 20 participants and will meet weekly for 2 hours. By the end of the program, participants will be encouraged to create a personalized action plan focusing on exercise and other healthy lifestyle choices.
  Other Names: Support group; Psychoeducation; Exercise support; Self-care

SUMMARY:
The purpose of this study is to pilot-test a culturally-tailored, community-based educational program for African-Americans, focusing on how to use exercise and other self-management strategies to reduce depressive symptoms and improve health. This study will explore what type of additional support would encourage depressed African-Americans to exercise regularly. The investigators hypothesize that participants will report greater frequency of exercise and lower depression scores at the end of the program than they did at baseline. However, this study is not adequately powered to test this hypothesis - the main goal is to assess feasibility, acceptability and satisfaction of the pilot intervention.

DETAILED DESCRIPTION:
Several studies have documented the effectiveness of exercise as a treatment for depression. However, these studies have used supervised exercise in medical school or university environments and have included mostly middle-class White populations. Little is known regarding how to translate these findings to real world settings or to minority populations. Exercise may be a particularly beneficial option for African-Americans suffering from depression. African-Americans face significant disparities in depression care. At least a part of these disparities are due to lack of trust in the healthcare system and negative attitudes toward antidepressants. Our goal is to pilot-test a culturally-tailored, community-based exercise support program for depressed African-Americans. We will recruit participants who screened positive for moderate depressive symptoms when they enrolled in the African-American Health Coalition's Free Exercise Card Program, but who are exercising less than 3 times per week. They will participate in a 6-week educational self-care group focusing on how to use exercise and other self-help tools to reduce depressive symptoms. Participants will be encouraged to create action plans regarding exercise and other healthy lifestyle changes. Groups will also provide culturally-tailored information about depression therapies, such as antidepressants and psychotherapy, and discuss strategies for obtaining quality health care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* African-American or of African-American descent
* Currently participating in the African-American Health Coalition Free Exercise-Card Program
* Experiencing moderate depressive symptoms, as indicated by a score of 10-20 on the Depression Scale of the Patient Health Questionnaire (PHQ-9.
* Exercising less than three times per week (for a minimum of 30 minutes per session) over the past month

Exclusion Criteria:

* Actively suicidal
* If a health care provider, AAHC staff member, or an investigator feel that participation in the program may endanger the participant's health or safety.
* Known mental or cognitive impairments
* Known condition that precludes their ability to feasibly participate in a support group session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in depression severity, as measured by the Depression Scale of the Patient Health Questionnaire (PHQ-9) | Week 1 (pre-test) and week 6 (post-test)

SECONDARY OUTCOMES:
Frequency of exercise using the International Physical Activity questionnaire(IPAQ). | Week 1 and Week 6
Attitudes about exercise, exercise self-efficacy and readiness to exercise using physical activity assessment scale (PAAS). | Week 1 and Week 6
Use of guideline-concordant depression therapies | week 1 and week 6
Acceptability of antidepressant therapy and counseling | week 1 and week 6
Depression self-care behaviors | week 1 and week 6
Satisfaction with program | week 6
Attendance to sessions | Each week for 6 weeks
Depression care self-efficacy | week 1 and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Nicolaidis, MD,MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- African American Health Coalition, Portland, Oregon, United States